CLINICAL TRIAL: NCT06481917
Title: Feasibility and Effectiveness of a Specialized Home-based Nurse Intervention on the Completion of Advance Care Plans of Patients at High Risk of Death After Discharge From Acute Care Geriatric Departement
Brief Title: Home-based Nurse Intervention in the Care of High Risk of Death Patients After Discharge From Geriatric Department
Acronym: SAPHARI
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Lille Catholic University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: RC-P00119
Record Dates: First submitted 2024-06-25; First posted 2024-07-01 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-07

CONDITIONS: Health Services for the Aged; Advance Care Planning
Keywords: Elderly; Advance care plan; DAMAGE score; High risk of mortality; Discharge from acute care geriatric department

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Advance care plan (Experimental): Scheduling of 2 home visits by an expert nurse in the month following the return home and proposal to carry out an advance care plan.
  Interventions: Other: Advance care plan; Other: Ergonomic analysis; Other: Evaluation of intervention acceptability
- Usual care (No Intervention): Usual care with the possibility of proposing ACP according to the department's habits

INTERVENTIONS:
Other: Advance care plan — Scheduling of 2 home visits by an expert nurse in the month following the return home and proposal to carry out an advance care plan.
  Arms: Advance care plan
Other: Ergonomic analysis — Ergonomic analysis throughout the intervention
  Arms: Advance care plan
Other: Evaluation of intervention acceptability — Evaluation of intervention acceptability after each home visit with patients and caregivers using a questionnaire
  Arms: Advance care plan

SUMMARY:
This study consists to evaluate the feasibility of a case-management intervention of Advance Care Plan (ACP) placement for elderly patients at high risk of death at twelve months discharged alive from acute geriatric medicine.

Feasibility will include the following indicators: rate of patients included and randomized, rate of patients remaining in the study, ACP rates achieved at one month.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 75 or over.
* Affiliated to a social security scheme.
* Hospitalized in an acute care geriatric department
* Discharged from hospital to home or residential facilities for dependent elderly people
* Targeted pathology or at least one incurable disease.
* At high risk of death in the twelve months following discharge according to the DAMAGE prognostic score (high-risk score group). A high risk of death is defined by a DAMAGE score > 50%.
* Rockwood Clinical frailty scale score greater than or equal to 7 at one month.

Exclusion Criteria:

* Refusal to participate in the study expressed by the patient or his/her legal representative, if applicable.
* Patients transferred to another Medicine-Surgery-Obstetrics department (only "medicine or surgery" in the elderly).
* Patients transferred to follow-up care and rehabilitation, palliative care, or returning home in palliative care.
* Patients who have already drawn up advance directives, chosen a trusted support person or discussed their end-of-life wishes with their doctor.
* Patients with proven severe neuro-cognitive disorders (in the medical record with a Mini-Mental State Examination (MMSE) score below 10 or in the absence of knowledge of the degree of severity and/or a recent previous MMSE score taken in a stable period, the referring practitioner, a geriatrician with expertise in this field, will assess whether the patient is unfit to state his or her advance directives at the time of inclusion.

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 104 (Estimated)
Dates: Start 2024-10 (Estimated); Primary Completion 2026-05 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
Rate of included patients | 12 months
Rate of patients remaining in the study | 12 months
Advance care planning rate achieved | 12 months

SECONDARY OUTCOMES:
Rate of compliance to advance directives | 12 months
  Rate of compliance with the patient's advance directives one year after discharge from hospital; compliance to the the following situations will be identified:
  * The patient is still alive: wishes to be re-hospitalized / does not wish to be re-hospitalized / has not made a decision.
  * The patient is deceased: place of death specified: hospital, home or other / no decision taken.
Hospital Anxiety and Depression Scale (HADS) of caregivers and carers | 12 months
  Anxiety-depressive symptomatology of caregivers will be assessed using the Hospital Anxiety and Depression Scale (HADS) in the event of patient death, if this occurs within one year of discharge from hospital. The HAD scale is a screening instrument for anxiety and depressive disorders. It comprises 14 items rated from 0 to 3. Seven questions relate to anxiety (total A) and seven to depression (total D), giving two scores (maximum score for each = 21). To screen for anxiety and depressive symptoms, the following interpretation can be proposed for each of the scores (A and D) each of the scores (A and D):
  * 7 or less: no symptoms
  * 8 to 10: doubtful symptomatology - 11 or more: definite symptomatology.
Questionnaire to evaluate the acceptability of the intervention | 12 months
  The acceptability of the intervention will be assessed by a questionnaire after each home visit at 7 days and one month, with patients and caregivers in the intervention group.
EQ-5D-3L scale score | 12 months
  Changes in the quality of life of patients and caregivers one month after hospital discharge will be measured by changes in the EQ-5D-3L scale score. EQ-5D is a standardised measure of health-related quality of life.n EQ-5D-3L, the five dimensions each have three response levels of severity.
  Respondents are asked to choose the statement in each dimension that best describes their health status on the day they are surveyed. Their responses are coded as a number (1, 2, or 3) that corresponds to the respective level of severity: 1 indicates no problems, 2 some problems, and 3 extreme problems. In this way, a person's health state profile can be defined by a 5-digit number, ranging from 11111 (having no problems in any of the dimensions) to 33333 (having extreme problems in all the dimensions).

CONTACTS AND LOCATIONS:
Overall Officials: Fabien VISADE, Principal Investigator — Hôpital Saint Philibert, GHICL
Locations (6):
- France (6):
  - CHU d'Amiens, Amiens
  - CHU de Caen, Caen
  - CHU de Lille, Lille
  - Hôpital Saint Vincent de Paul (GHICL), Lille
  - Hôpital Saint-Philibert (GHICL), Lomme
  - CHU de Rouen, Rouen

IPD SHARING:
Plan to Share IPD: No